CLINICAL TRIAL: NCT02638662
Title: Does Stress Affect In-Vitro Fertilization (IVF) Outcome?
Brief Title: Stress Level and the Relationship With IVF Outcomes.
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0903010295
Record Dates: First submitted 2015-10-06; First posted 2015-12-23 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- First time IVF patients. Observational: Those who are doing IVF for the first time.
  Interventions: Other: Observational
- Donors Observational: Those who are doing IVF for the sole purpose of donating their eggs.
  Interventions: Other: Observational
- 2 or more IVF cycles Obervational: Those who have done IVF 2 or more times with no success.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Questionnaires are completed such as self-evaluation questionnaire (STAI), Beck Depression Inventory, FertiQol International and Daily stress questionnaire

SUMMARY:
The effect of stress on IVF outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to describe the pattern of psychological distress (depression, anxiety and stress) as assessed by both subjective and objective measures throughout the course of IVF treatment and to investigate its impact on IVF outcome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women undergoing IVF at CRMI Ages 20-44

Patients will be divided in different groups depending on whether:

1. They are donating oocytes (control group).
2. They are undergoing IVF for the first time.
3. They are undergoing IVF for the third time and have either failed or succeeded the prior time.

Exclusion Criteria:

* Any patients who are not candidates for IVF
* Any women who have any past or current medical condition unrelated to their infertility concurrent to their history of infertility (e.g., gastrointestinal disease)

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: IVF patients doing IVF for the first time, or doing it for the third or more time doing it for the sole purpose to donate their eggs
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Biomarkers Cortisol and adrenocorticotropic hormone ACTH. | 28-35 days

SECONDARY OUTCOMES:
Questionnaires to be completed are Life Orientation Test-R | 28-35 days
Self- Evaluation Questionnaire (STAI) | 28-35 days
  Questionnaire
FertiQOL International | 28-35 days
Beck Depression Inventory | 28-35 days
  Questionnaire
Daily Stress Questionnaire | 28-35 days
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steven Spandorfer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No